CLINICAL TRIAL: NCT07028684
Title: Effects of Foot Reflexology Massage in Pain, Sleep and Quality of Life in Females With Migraine
Brief Title: Effects of Foot Reflexology Massage in Migraine
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karabuk University (Other)
Responsible Party: Principal Investigator, Tarik Ozmen, Professor, Karabuk University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KBU-FTR-2025-2178
Record Dates: First submitted 2025-06-11; First posted 2025-06-19 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-06

CONDITIONS: Migraine Disease
Keywords: Migraine; Massage; Headache
MeSH Terms: conditions — Migraine Disorders; Headache | interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Intervention Model Description: The study includes two groups with massage and control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): No treatment other than medication will be given for migraine.
- Experimental (Experimental): Reflexology massage will be applied twice a week for 30 minutes per session, for a total of 10 sessions.
  Interventions: Other: Reflexology Massage

INTERVENTIONS:
Other: Reflexology Massage — Reflexology massage will be applied twice a week for 30 minutes per session, for a total of 10 sessions. The treatment will begin by relaxing the ankle with a few passive movements. Reflexology massage will be applied to the right foot first and then to the left foot.
  Target Areas to be Applied to the Right Foot: Brain, Pineal, Hypophysis, Hypothalamus and Thalamus, Temples, Eye area and Optic nerve, Ear area, Middle ear and Balance point, Neck.
  Other areas to be applied to the right foot: Thyroid and Parathyroid, Lung, Liver, Face area, Speech center and Thymus, Teeth, Diaphragm, Vertebra, Extremities.
  Areas to be applied to the left foot: Kidney, Diaphragm, Intestines, Neck, Vertebra, Extremities.
  The session is completed from the left foot by applying to the lymph inlet, lymph channel and diaphragm from both feet.
  Arms: Experimental

SUMMARY:
Migraine is a primary headache type that usually manifests itself with unilateral, moderate to severe throbbing headaches, often accompanied by symptoms such as nausea, vomiting, and sensitivity to light and sound. The prevalence and impact of headaches are more pronounced, especially among women, and this condition is among the top five causes of disability in women. Reflexology, one of the complementary treatment methods, is an alternative medical practice that produces beneficial effects on the human body by applying pressure to specific points or areas called "reflex areas" on the feet, hands, and ears.The aim of this randomized controlled trial was to evaluate the effects of foot reflexology massage on pain, sleep, and quality of life in women with migraine. All patients included in this study will be evaluated with the following tests and scales three times: before, after, and 2 weeks after the end of the 5-week (10 sessions in total) treatment. After the initial evaluations of the study, migraine patients will be divided into 2 groups using a simple random sampling method in the computer randomization program. The first group will receive a foot reflexology massage. The second group will be the control group.

DETAILED DESCRIPTION:
Migraine is a primary headache type that usually manifests itself with unilateral, moderate to severe throbbing headaches, often accompanied by symptoms such as nausea, vomiting, and sensitivity to light and sound. The prevalence and impact of headaches are more pronounced, especially among women, and this condition is among the top five causes of disability in women. Reflexology, one of the complementary treatment methods, is an alternative medical practice that produces beneficial effects on the human body by applying pressure to specific points or areas called "reflex areas" on the feet, hands, and ears. Reflexology can be used as a complementary or supportive method of treatment because it is a massage form that regulates complex body functions and has relaxing and loosening effects. In studies; It has been found that foot reflexology reduces patients' pain and improves their sleep quality. The aim of this randomized controlled trial was to evaluate the effects of foot reflexology massage on pain, sleep, and quality of life in women with migraine. All patients included in this study will be evaluated with the following tests and scales three times: before, after, and 2 weeks after the end of the 5-week (10 sessions in total) treatment. After the initial evaluations of the study, migraine patients will be divided into 2 groups using a simple random sampling method in the computer randomization program. The first group will receive a foot reflexology massage. The second group will be the control group.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-45
* Being diagnosed with migraine by a neurologist according to the International Headache Society (IHS) criteria
* Volunteering to participate in the study
* Being able to read and write
* Not having entered menopause

Exclusion Criteria:

* Any neurological or musculoskeletal disease other than migraine
* History of cervical or cranial surgery
* Irritation or ulceration on the skin area to be reflexologized
* Receiving non-drug migraine treatment (acupuncture, dry needle, etc.)
* Those who have received physiotherapy at least 6 months ago
* Presence of diabetic foot
* Open wounds on the foot
* Pregnant individuals or individuals who become pregnant during the study

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2025-10-15 (Estimated); Study Completion 2025-10-15 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale | 5 weeks
  Pain intensity will be assessed with a visual analog scale. The patient marks his/her own pain on a 10 (represents "worst pain imaginable") cm ruler with painlessness 0 (represents "no pain") at one end and the most severe pain possible at the other end.

SECONDARY OUTCOMES:
Headache Impact Test | Five weeks
  It will be used to measure the impact of headache on participants' quality of life. Items in this test assess areas such as vitality, pain and psychological distress, as well as sociability, role and cognitive functioning. Each item is answered on a 5-point Likert scale. The final score is determined by summing the scores on the six items, ranging from 36 to 78 points, with a higher score indicating a greater effect.
Pittsburgh Sleep Quality Index | Five weeks
  Sleep quality will be assessed with a scale consisting of 24 questions and 7 categories. Each item is evaluated with a score between 0 and 3, with 0 being no problems and 3 being serious problems. The total score is between 0-21. A high total score indicates poor sleep quality.
Migraine disability assessment | Five weeks
  It is a questionnaire that has proven to be reliable and valid in determining the degree of disability caused by migraine. MIDAS assesses the degree of disability from 1 to 4 based on the number of days (score). Grade I: Little or no disability (0-5 days), Grade II: Mild disability (6-10 days), Grade III: Moderate disability (11-20 days) and Grade IV (21+ days): Indicates severe disability.
24-h Migraine Quality of Life Questionnaire | Five weeks
  The 24-hour quality of life scale will be used to evaluate the changes in the quality of life of the patients within 24 hours after the first dose of migraine medication. The scale has 3 sections and a total of 15 items covering quality of life areas under the headings of Migraine symptoms, Emotions, Worries, Work Functionality, Social Functionality, Energy-Vitality. The total score is minimum 15 and maximum 105. The higher the scores the individual receives from the scale, the higher the quality of life of the individual, and the lower the score, the lower the quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Karabuk University, Karabük, Turkey (Türkiye)